CLINICAL TRIAL: NCT00809510
Title: A Study of the Long-term Safety of ABT-089 for Subjects With Mild-to-moderate Alzheimer's Disease Who Participated in the M06-876 Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-745
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — pozanicline

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABT-089

INTERVENTIONS:
Drug: ABT-089 — 20 mg ABT-089 taken once-daily for 6 months

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of ABT-089 in adults with mild-to-moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* The subject was randomized into Study M06-876 and completed the study.
* The subject must remain on the same dose of AChEI that was used during the M06-876 study.
* The subject is in general good health, as judged by the investigator

Exclusion Criteria:

* The subject is currently, or plans to participate in another experimental study during the course of this trial.
* The subject anticipates a move outside the geographic area of the investigative site or is planning extended travel inconsistent with the recommended visit intervals.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety Assessments (i.e., ECG, clinical laboratory tests, vital signs, weight, AE assessment, physical and brief neurological examinations) | Month 1, 2, 4, 6

SECONDARY OUTCOMES:
ADAS-Cog, CIBIC-plus, MMSE, QoL-AD | Month 1, 2, 4, 6

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lenz, Study Director — Abbott
Locations (22):
- United States (22):
  - Site Reference ID/Investigator# 16543, Phoenix, Arizona
  - Site Reference ID/Investigator# 16528, Sun City, Arizona
  - Site Reference ID/Investigator# 16524, Fresno, California
  - Site Reference ID/Investigator# 16520, San Diego, California
  - Site Reference ID/Investigator# 16521, Santa Monica, California
  - Site Reference ID/Investigator# 16533, Hamden, Connecticut
  - Site Reference ID/Investigator# 16516, Brooksville, Florida
  - Site Reference ID/Investigator# 16510, Deerfield Beach, Florida
  - Site Reference ID/Investigator# 16508, Delray Beach, Florida
  - Site Reference ID/Investigator# 16515, Miami, Florida
  - Site Reference ID/Investigator# 16545, Palm Beach Gardens, Florida
  - Site Reference ID/Investigator# 16541, Sunrise, Florida
  - Site Reference ID/Investigator# 16542, Tampa, Florida
  - Site Reference ID/Investigator# 16529, West Palm Beach, Florida
  - Site Reference ID/Investigator# 16526, Indianapolis, Indiana
  - Site Reference ID/Investigator# 16527, Eatontown, New Jersey
  - Site Reference ID/Investigator# 16523, Ridgewood, New Jersey
  - Site Reference ID/Investigator# 16532, New York, New York
  - Site Reference ID/Investigator# 16519, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 16525, Centerville, Ohio
  - Site Reference ID/Investigator# 16507, Wichita Falls, Texas
  - Site Reference ID/Investigator# 16509, Bennington, Vermont